CLINICAL TRIAL: NCT02741999
Title: A Diagnostic Screening Trial Seeking AL Amyloidosis Very Early
Acronym: SAVE
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12016
Record Dates: First submitted 2016-04-11; First posted 2016-04-18 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Plasma Cell Dyscrasia; Monoclonal Gammopathy
MeSH Terms: conditions — Paraproteinemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow and peripheral blood samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol seeks to enroll smoldering multiple myeloma (SMM) and monoclonal gammopathy of undetermined significant (MGUS) patients with λ light chain (LC) involvement, a group of patients for whom standard of care is observation not treatment. Patients with SMM and MGUS have a precursor plasma cell disorder from which light chain amyloidosis (AL) can evolve. In this trial, enrolled subjects will have blood and if available bone marrow cells evaluated by molecular testing to determine their clonal λ LC variable region (VL) germline gene. Seventy percent of AL cases involve just 7 germline donors, 5 of which are λ germline donors. The hypothesis that will be tested with this protocol is that the presence of AL germline genes associated with AL in patients with a pre-existing diagnosis of λ SMM or λ MGUS indicates the presence of AL or risk of progression to AL.

DETAILED DESCRIPTION:
In this trial up to 200 patients with either λ light chain (LC) monoclonal gammopathy of undetermined significance (MGUS) or λ LC smoldering multiple myeloma (SMM) with a κ::λ LC ratio < 0.26 and whose λ minus κ LC difference (dFLC) is greater than 23 mg/L will be recruited. Heavy chain type will not affect patient eligibility as long as the involved LC is λ type.

Patients may learn about the trial through internet advertisements and contact the data manager to receive the study's enrollment documents. Patient recruitment will be open to all eligible patient within the United States. Informed consent may be obtained in person or by phone. After the patient has completed a HIPPA release form, the patient's physician will be contacted and informed of the patient's consent to this study and will be asked to provide medical records for screening. If the patient is found eligible, the patient and physician will be informed of the required samples for the protocol, which include peripheral blood and marrow aspirate, if available, with both taken during routine clinical procedures. Prepaid FedEx boxes will be provided by the study to ship research samples to Tufts Medical Center for remote patients.

Both the peripheral blood and marrow samples will be tested for the presence of variable region (VL) germline genes in our Tufts Medical Center laboratory. In addition, plasma isolated from the peripheral blood sample (as well as the corresponding identified germline gene) will be sent to the laboratory of Dr. Jonathan Wall at the University of Tennessee for assay analysis. The assay will seek to distinguish the presence of amyloidogenic vs. non-amyloidogenic light chains. Germline gene results from Tufts Medical Center will be shared with patients and their physicians; however, University of Tennessee assay analysis will not be shared due to its experimental nature.

The analysis of this trial will be based on the frequency with which enrolled MGUS and SMM patients are found to have genes associated with light chain amyloidosis (AL), are found to have asymptomatic AL or symptomatic AL, or progress to AL. The diagnosis of AL is a tissue diagnosis. If amyloidosis is suspected at any time during a subject's participation, their physician will be contacted and given recommendations regarding diagnostic tests and disease staging.

ELIGIBILITY:
Inclusion Criteria:

* MGUS and SMM patients with λ LC involvement with dFLC > 23 mg/L and κ:: λ free LC ratios < 0.26. Subjects must be able to share their medical records and ship us bone marrow and blood samples.

Exclusion Criteria:

* MGUS and SMM patients with light chains that do not meet the inclusion criteria as well as patients with κ LC involvement or active myeloma will not be included. And patients who are unable to send us blood and marrow for any reason will not be eligible.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll up to 200 MGUS and SMM patients with λ LC involvement with dFLC >23 mg/L and κ:: λ free LC ratio <0.26. Subjects must be able to share their medical records and ship bone marrow and blood samples to our laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
Observation of disease progression in participants with AL-associated VL germline genes | 5 years
  After sequencing of their light chain (LC) variable region (VL) germline gene, subjects with light chain amyloidosis (AL) associated sequences will be followed for up to 5 years to monitor the potential progression of their disease to AL amyloidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Comenzo, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bodi K, Prokaeva T, Spencer B, Eberhard M, Connors LH, Seldin DC. AL-Base: a visual platform analysis tool for the study of amyloidogenic immunoglobulin light chain sequences. Amyloid. 2009 Mar;16(1):1-8. doi: 10.1080/13506120802676781. PMID 19291508
- [Background] Comenzo RL, Wally J, Kica G, Murray J, Ericsson T, Skinner M, Zhang Y. Clonal immunoglobulin light chain variable region germline gene use in AL amyloidosis: association with dominant amyloid-related organ involvement and survival after stem cell transplantation. Br J Haematol. 1999 Sep;106(3):744-51. doi: 10.1046/j.1365-2141.1999.01591.x. PMID 10468868
- [Background] Comenzo RL, Zhang Y, Martinez C, Osman K, Herrera GA. The tropism of organ involvement in primary systemic amyloidosis: contributions of Ig V(L) germ line gene use and clonal plasma cell burden. Blood. 2001 Aug 1;98(3):714-20. doi: 10.1182/blood.v98.3.714. PMID 11468171
- [Background] Chaulagain CP, Comenzo RL. How we treat systemic light-chain amyloidosis. Clin Adv Hematol Oncol. 2015 May;13(5):315-24. PMID 26352777
- [Background] Dasari S, Theis JD, Vrana JA, Meureta OM, Quint PS, Muppa P, Zenka RM, Tschumper RC, Jelinek DF, Davila JI, Sarangi V, Kurtin PJ, Dogan A. Proteomic detection of immunoglobulin light chain variable region peptides from amyloidosis patient biopsies. J Proteome Res. 2015 Apr 3;14(4):1957-67. doi: 10.1021/acs.jproteome.5b00015. Epub 2015 Mar 20. PMID 25734799
- [Background] Dispenzieri A, Kyle RA, Katzmann JA, Therneau TM, Larson D, Benson J, Clark RJ, Melton LJ 3rd, Gertz MA, Kumar SK, Fonseca R, Jelinek DF, Rajkumar SV. Immunoglobulin free light chain ratio is an independent risk factor for progression of smoldering (asymptomatic) multiple myeloma. Blood. 2008 Jan 15;111(2):785-9. doi: 10.1182/blood-2007-08-108357. Epub 2007 Oct 17. PMID 17942755
- [Background] Dubrey SW, Cha K, Anderson J, Chamarthi B, Reisinger J, Skinner M, Falk RH. The clinical features of immunoglobulin light-chain (AL) amyloidosis with heart involvement. QJM. 1998 Feb;91(2):141-57. doi: 10.1093/qjmed/91.2.141. PMID 9578896
- [Background] Kourelis TV, Kumar SK, Go RS, Kapoor P, Kyle RA, Buadi FK, Gertz MA, Lacy MQ, Hayman SR, Leung N, Dingli D, Lust JA, Lin Y, Zeldenrust SR, Rajkumar SV, Dispenzieri A. Immunoglobulin light chain amyloidosis is diagnosed late in patients with preexisting plasma cell dyscrasias. Am J Hematol. 2014 Nov;89(11):1051-4. doi: 10.1002/ajh.23827. Epub 2014 Sep 2. PMID 25111004
- [Background] Kyle RA, Rajkumar SV. Monoclonal gammopathy of undetermined significance and smoldering multiple myeloma. Curr Hematol Malig Rep. 2010 Apr;5(2):62-9. doi: 10.1007/s11899-010-0047-9. PMID 20425398
- [Background] Kyle RA, Remstein ED, Therneau TM, Dispenzieri A, Kurtin PJ, Hodnefield JM, Larson DR, Plevak MF, Jelinek DF, Fonseca R, Melton LJ 3rd, Rajkumar SV. Clinical course and prognosis of smoldering (asymptomatic) multiple myeloma. N Engl J Med. 2007 Jun 21;356(25):2582-90. doi: 10.1056/NEJMoa070389. PMID 17582068
- [Background] Larsen JT, Kumar SK, Dispenzieri A, Kyle RA, Katzmann JA, Rajkumar SV. Serum free light chain ratio as a biomarker for high-risk smoldering multiple myeloma. Leukemia. 2013 Apr;27(4):941-6. doi: 10.1038/leu.2012.296. Epub 2012 Oct 16. PMID 23183428
- [Background] Perfetti V, Casarini S, Palladini G, Vignarelli MC, Klersy C, Diegoli M, Ascari E, Merlini G. Analysis of V(lambda)-J(lambda) expression in plasma cells from primary (AL) amyloidosis and normal bone marrow identifies 3r (lambdaIII) as a new amyloid-associated germline gene segment. Blood. 2002 Aug 1;100(3):948-53. doi: 10.1182/blood-2002-01-0114. PMID 12130507
- [Background] Perfetti V, Palladini G, Casarini S, Navazza V, Rognoni P, Obici L, Invernizzi R, Perlini S, Klersy C, Merlini G. The repertoire of lambda light chains causing predominant amyloid heart involvement and identification of a preferentially involved germline gene, IGLV1-44. Blood. 2012 Jan 5;119(1):144-50. doi: 10.1182/blood-2011-05-355784. Epub 2011 Nov 8. PMID 22067386
- [Background] Rajkumar SV, Kyle RA, Therneau TM, Melton LJ 3rd, Bradwell AR, Clark RJ, Larson DR, Plevak MF, Dispenzieri A, Katzmann JA. Serum free light chain ratio is an independent risk factor for progression in monoclonal gammopathy of undetermined significance. Blood. 2005 Aug 1;106(3):812-7. doi: 10.1182/blood-2005-03-1038. Epub 2005 Apr 26. PMID 15855274
- [Background] Zhou P, Comenzo RL, Olshen AB, Bonvini E, Koenig S, Maslak PG, Fleisher M, Hoffman J, Jhanwar S, Young JW, Nimer SD, Boruchov AM. CD32B is highly expressed on clonal plasma cells from patients with systemic light-chain amyloidosis and provides a target for monoclonal antibody-based therapy. Blood. 2008 Apr 1;111(7):3403-6. doi: 10.1182/blood-2007-11-125526. Epub 2008 Jan 23. PMID 18216299
- [Background] Zhou P, Hoffman J, Landau H, Hassoun H, Iyer L, Comenzo RL. Clonal plasma cell pathophysiology and clinical features of disease are linked to clonal plasma cell expression of cyclin D1 in systemic light-chain amyloidosis. Clin Lymphoma Myeloma Leuk. 2012 Feb;12(1):49-58. doi: 10.1016/j.clml.2011.09.217. Epub 2011 Nov 18. PMID 22100494
- [Background] Zhou P, Ma X, Iyer L, Chaulagain C, Comenzo RL. One siRNA pool targeting the lambda constant region stops lambda light-chain production and causes terminal endoplasmic reticulum stress. Blood. 2014 May 29;123(22):3440-51. doi: 10.1182/blood-2013-10-535187. Epub 2014 Apr 10. PMID 24723680